CLINICAL TRIAL: NCT04729179
Title: Cannabidiol for Fibromyalgia -The CANNFIB Trial Protocol for a Randomized, Double-blind, Placebo-controlled, Parallel-group, Single-center Trial
Brief Title: Cannabidiol for Fibromyalgia (The CANNFIB Trial)
Acronym: CANNFIB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P142; 2019-002394-59 (EudraCT Number); H-20047715 (Other: Regional Ethical Committee Journal Number)
Record Dates: First submitted 2021-01-18; First posted 2021-01-28 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Fibromyalgia
Keywords: Cannabidiol; Chronic widespread pain; Sleep disturbances; Fatigue; Functional ability; Quality of life
MeSH Terms: conditions — Fibromyalgia; Chronic Pain; Parasomnias; Fatigue | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, parallel-group, single center trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The project medication is manufactured specifically for research purposes, and the cannabidiol and cannabidiol placebo pills are identical in appearance, taste, and smell. The cannabidiol and placebo tablet packages are labelled with a unique Dispensing Unit Number (DUN). It is concealed to all involved parties (the participant, care provider, investigator qand outcomes assessor), but the database manager, wether the DUN can be identified as cannabidiol package or a placebo package.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (Experimental): Participants will start with 10 mg of cannabidiol daily and the dose will be escalated every third day until the maximum dosage of 50 mg is reached (after two weeks). The participants be on the 50 mg dosage of cannabidiol for 24 weeks.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): Placebo is administered as tablets of 10 mg that are identical in appearance, taste, and smell to the Cannabidiol tablets.The participants will be on the 50 mg dosage of placebo for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — Participants will start with 10 mg of cannabidiol daily and the dose will be escalated every third day until the maximum dosage of 50 mg is reached (after two weeks). The participants be on the 50 mg dosage of cannabidiol for 24 weeks.
  Other Names: Cannabidiol active ingredient
  Arms: Cannabidiol
Drug: Placebo — Placebo is administered as tablets of 10 mg that are identical in appearance, taste, and smell to the Cannabidiol tablets.The participants will be on the 50 mg dosage of placebo for 24 weeks.
  Other Names: Cannabidiol Placebo
  Arms: Placebo

SUMMARY:
Fibromyalgia is serious chronic pain condition which is often accompanied by sleep disturbances, fatigue and disability and reduced quality of life. There is no cure and treatments are based on reliving symptoms and maintaining function. The currently available medical treatments are not helping many patients, and many get side-effects. Medical cannabis is sought after among patients and many use this medication un-licenced, although it is not properly documented if it works or is safe. Therefore, it is necessary to investigate the effects and safety of medical cannabis in a properly designed randomized trial. The aim of the study is to investigate if cannabidiol (CBD) can improve pain, sleep, function and quality of life in patients with fibromyalgia. The study will include 200 patients, who will receive either cannabidiol or placebo over a period of 24 weeks. Participants will be closely looked after for improvements in their condition and for potential side-effects to ensure safety.

DETAILED DESCRIPTION:
BACKGROUND: Fibromyalgia is a serious chronic pain condition affecting 2-5 % of the background population. The disease burden in most affected individuals is substantial; with widespread musculoskeletal pain, high pain intensity, often accompanied by sleep disturbances, fatigue, cognitive dysfunction, and emotional distress. Fibromyalgia is associated with disability and muscle fatigue, affecting daily life activities, leading to poor social participation and incapacity for normal employment. Studies have shown that many patients, are not satisfied with the treatments offered, and rate their health and quality of life after treatment as poor.

There is currently is no cure for fibromyalgia, and management aiming at symptom reduction and maintenance of optimal functioning is recommended by clinical guidelines, including both non-pharmacological and pharmacological treatment strategies. Recommendations for the pharmacological treatment of fibromyalgia propose antidepressants and anticonvulsants, which target central pain processing mechanisms. These treatments have been tested in controlled trials for their efficacy in patients with fibromyalgia, and meta-analyses on these interventions have revealed that overall effect sizes are modest, as only a minority of patients have substantial benefit (patient reported pain relief of 50% or greater), while more have moderate benefit (patient reported pain relief of 30% or greater). Many patients have no or minimal benefit or will discontinue the treatment due to side effects. However, it appears that even moderate reductions in pain may lead to considerable increase in self-reported quality of life and other outcome domains in this specific patient population.

Medical cannabis is popularly advocated for different health conditions including chronic pain, both among politicians and in the general population in Denmark, although evidence is sparse efficacy and on what types of medical cannabis to use and what dosages to prescribe for the different conditions. In addition, safety issues such as adverse events and serious adverse events is not properly assesed. Physicians are reluctant to prescribe medical cannabis to their patients, and many patients living with chronic pain are known to self-administer unlicensed medical cannabis. The extent of actual cannabis use is unknown, although, one study has documented that 13% of patients with fibromyalgia use cannabis regularly with a more extensive use among male patients compared to females. Numbers from a Danish context show that only 17 out of 286 (6%), patients with fibromyalgia participating in a multidisciplinary rehabilitation program in Bispebjerg and Frederiksberg hospital during 2018, stated that they were using self-administrated cannabis on a regular basis (unpublished data). As self-administrated off-label use of cannabis is illegal in Denmark, this number may well be underreported. Still, individuals diagnosed with fibromyalgia who do admit to cannabis use, are sharing stories with health professionals about how unlicensed cannabis has improved their coping with everyday life, functional ability, pain, sleep, fatigue, mood and overall health related quality of life. Such compelling stories cannot be ignored and underline the necessity of exploring the efficacy of medical cannabis in a proper research design (i.e. with good internal validity).

The use of the cannabis plant for medical purposes is limited in Europe and the European addiction societies stresses the need for further studies on the efficacy and possible dangers regarding medical cannabis intake. Regulations are lacking on registration and medical indications, and the development of uniform compounds regarding strength and types of products and rules concerning sales and marketing.

In Denmark, production and distribution of medical cannabis is illegal. However, starting from January 1st, 2018, a four-year pilot scheme has been legalized and approved by the Danish Medicines Agency, allowing for medical cannabis in the treatment of conditions such as multiple sclerosis, spinal injuries and nausea after chemotherapy and neuropathic pain. Although patients suffering from fibromyalgia have few treatment options for management of their disabling condition, this group is not included in the pilot scheme. However, it is legal for physicians to prescribe cannabis for this and other patient groups.

Medical cannabis Medical cannabis is the term for medications derived from dried cannabis plants in the form of capsules, pills or extracts/oils. The top shoot of the plant contains 100 cannabinoids that are divided into two subgroups; Delta-9-tetrahydrocannabinol (THC) and cannabidiol (CBD), affecting the cannabinoid type 1 receptors located in the central nervous system, and the cannabinoid type 2 receptors located outside of the central nervous system. While the THC cannabinoids have psychoactive, appetite stimulating and nausea reducing effects, cannabidiol has anti-inflammatory, anti-convulsive and immune modulating effects. Studies are inconclusive regarding the effect of cannabidiol on appetite and food intake. Cannabinoids are known to be highly lipophilic and to accumulate in fatty tissue, and may influence the metabolism, fat distribution and accumulation in users. It has been implicated that both TCH and CBD have pain reducing effects. CBD is confirmed to have a favorable safety profile compared to THC.

The US Food and Drug Administration (FDA), has approved Epydiolex® as the first prescription cannabis drug derived from the cannabis plant, for treating rare and severe forms of epilepsy. Synthetically manufactured cannabis such as dronabinol (USA) and nabilone (USA and UK), have been approved earlier in the treatment of nausea after chemotherapy. The only synthetic cannabis based approved drug in Denmark is Sativex® for the treatment of multiple sclerosis. However, none of the cannabis drugs are currently approved for the treatment of chronic pain conditions.

Evidence is sparse on medical cannabis in the treatment of fibromyalgia. In a Cochrane review on herbal cannabis (hashish, marihuana), plant-based and synthetic cannabinoids for fibromyalgia, only two out of four identified studies on the topic were included, due to small sample sizes, short-term duration and poor reporting of the other studies. The two studies were both on synthetic cannabinoid (nabilone). No high-quality studies on plant-based cannabis could be identified. Evidence for efficacy was inconsistent as one study favored nabilone on pain and quality of life, compared to placebo, and the other study favored nabilone on sleep compared to Amitriptyline (anti-depressant). However, the quality of the studies was low, and tolerability was low due to side effects.

Recent systematic reviews, have investigated the existing evidence on the effectiveness of cannabinoids for chronic non-cancer pain, including fibromyalgia. No impact on physical and emotional functioning has been found, and only low-quality evidence found improved sleep and patient global impression of change. Thus, it was concluded to be unlikely that cannabinoids are effective in the treatment of non-cancer pain, as findings were inconsistent. Survey studies, however, have showed favorable effect on fibromyalgia symptoms and health-related quality of life, and improved pain management and sleep, among users of unlicensed cannabis compared to non-users, although no information on type and dosages of cannabis was given in the surveys. Negative patients' perspectives themes such as the high cost, the negative effects of cannabis and the "views of others", including their health care professionals, were also identified. A recent retrospective study showed significantly favorable outcomes on fibromyalgia symptoms among medical cannabis users, and only mild adverse events. However, the retrospective design, the relatively small sample size and short duration reduced the quality of the study.

Based on the high demand and an increasing popularity of medical cannabis - which is currently used unlicensed among many patients with fibromyalgia, despite the lack of high-quality evidence on efficacy and safety, a well-designed randomized trial with a large sample size and clinically relevant duration is warranted.

OBJECTIVES: The aim of this trial is to assess the efficacy and safety of cannabidiol use compared to placebo, and to evaluate the safety and tolerability of cannabidiol compared to placebo in patients with fibromyalgia over 24 weeks.

HYPOTHESES: The primary hypothesis of the study is that pain intensity will be significantly reduced in participants receiving cannabidiol compared to those receiving identically appearing placebo after 24 weeks.

Secondary hypotheses are that sleep quality and duration, activities of daily living and quality of life, will be improved in participants receiving cannabidiol compared to those receiving placebo after 24 weeks. It is also hypothesized that participants receiving cannabidiol will improve on several supportive exploratory secondary outcomes (see outcome measures section), and that a higher proportion of those receiving cannabidiol will have a substantial benefit (50 % pain reduction) and a moderate benefit (30 % pain reduction).

STUDY DESIGN: The trial is designed as a single-center, randomized, placebo-controlled, double blind and parallel-group trial.; the trial contains three periods: A pre-randomization screening period (week -8 to 0), a main trial period (week 0 to 24), and a post interventional observation period (week 24 to 36). The trial is designed to determine the efficacy and safety of cannabidiol use for patients with fibromyalgia.

The trial is scheduled to start inclusion of first patient first visit, February 2021 or as soon as possible thereafter, and the study period will go on for two year and end with the last patient last visit in December 2022.

Eligible participants, who are included at screening, will be randomized in a 1:1 manner to receive either cannabidiol 50 mg or placebo. Allocation will also be stratified based on sex (male vs. female), age and pain intensity (over vs. under 7 on the Fibromyalgia Impact Questionnaire Revised version (FIQ-R) pain numeric rating scale, to ensure that the groups are equal. A computer-generated randomization sequence will create subject identification numbers and allocate the subjects to treatment arms. The randomization sequence will be created by an independent biostatistician using a random number generator (SAS Proc Plan), and subsequently entered in the electronic Case Report Form (e-CRF), that will be developed specifically for the study, by an independent data manager. If unblinding of a participant is required due to an adverse event, the primary investigator can request to break the randomization code for the individual patient, via the independent data manager. The unblinding will always be performed at patient level and unblinding can take place any time during the day (24/7). Randomization and concealed allocation are done electronically in the e-CRF at the randomization visit (week 0).

The study will be conducted at the Parker Institute, Bispebjerg and Frederiksberg Hospital, University of Copenhagen. The Parker Institute is a well-established research institute and clinical department with secretariat, data managers and Good Clinical Practice (GCP) trained health care professionals including physicians and study nurses. Monitoring will be conducted from the initiation and throughout the trial by the GCP-unit at Bispebjerg and Frederiksberg hospital, in accordance with the GCP rules and regulations.

The trial will end when the last patient has completed the last visit as well as the 12-week post interventional observation period, or prematurely discontinued the intervention or withdrawn from the trial, which comes last.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Clinical diagnosis of fibromyalgia according to the American College of Rheumatology (ACR) 1990 criteria
* Average pain intensity ≥ 4 on a Numeric Rating Scale
* No use of medical cannabis (THC/CBD) within the last six months
* Proficiency in spoken Danish language and able to read and write in Danish

Exclusion Criteria:

* On-going participation in other medical trials for pain management of fibromyalgia
* Diagnosis of Rheumatoid Arthritis or other inflammatory diseases
* Diagnosis of other serious chronic diseases
* Impaired liver and kidney function
* Pregnancy or insufficient anti-conception therapy for fertile female participants
* Planning pregnancy or insufficient anti-conception use in fertile female partners of male participants
* Breast feeding
* Surgery scheduled for the trial period or within 3 months prior to enrollment
* History of or current diagnosis of cancer
* History of or current epilepsy and seizures
* History of or major depressive disorder
* History of a suicide attempt or any suicidal behavior
* A mental state that may impede compliance with the program
* History of severe psychiatric disorders
* History of or current cannabis abuse
* History of or current drug abuse
* History of or current alcohol abuse
* Severe personality disorder
* Current use of opioids, opioid antagonists (LDN) or similar strong analgesics
* Allergic reactions to the active ingredients in cannabidiol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

PRIMARY OUTCOMES:
Pain intensity | From baseline to week 24
  The primary endpoint is change in pain intensity, measured with the 0-10 pain numeric rating scale, from the Fibromyalgia Impact Questionnaire Revised. The minimum value is 0, which is the best outcome, indicating no pain. The maximum value is 10, which is the worst outcome, indicating the worst possible pain.

SECONDARY OUTCOMES:
Sleep quality | From baseline to week 24
  The first of six key secondary outcomes is change in sleep quality, measured with the Pittsburgh Sleep Quality Index; total score of overall sleep quality. Scores are ranging from 0 to 21, with lower scores indicating better sleep quality and higher scores indicating worse sleep quality.
Sleep duration | From baseline to week 24
  The second of six key secondary outcomes is change in sleep duration, measured with the Pittsburgh Sleep Quality Index; sleep duration domain, with number of hours of actual sleep during the night.
Objectively measured sleep duration | From baseline to week 24
  The third of six key secondary outcomes is change in objectively measured sleep duration, with number of hours of nightly sleep, measured with the Sens triaxial accelerometer device; MOTION® activity and sleep measurement system.
Objectively measured sleep patterns | From baseline to week 24
  The fourth of six key secondary outcomes is change in objectively measured sleep patterns, measured with the Sens triaxial accelerometer device; MOTION® activity and sleep measurement system, in which the different sleep phases during the night are indicated.
Activities of daily living | From baseline to week 24
  The fifth of six key secondary outcomes is change in Activities of Daily Living (ADL), measured with the Assessment of Motor and process skills (AMPS) test, which is an observation-based, standardized evaluation of the individual's ability to perform and complete activities of daily living. The measure is based on 16 ADL motor skills and 20 ADL process skills. Scores range from 0 to 4 on an ordinal scale, with 0 indicating the lowest level of ADL and 4 indicating the highest ADL level. Activities of daily living is also measured with the Activities of Daily Living Questionnaire, in which items are rated on a 4 point Likert scale from 0= no problem to 3=no longer able to complete the task. Scores are calculated for total and subscale scores and expressed as a percentage from 0 to 100%. Lower percentage indicates a higher ADL level, and higher percentage indicates a lower ADL level.
Health-related quality of life | From baseline to week 24
  The sixth of six key secondary outcomes is change in quality of life, measured with the EuroQol Self-Rated Health Questionnaire, developed by the EuroQual group and international network of multidisciplinary researchers.The scores goes from 0 -100, with 0 indicating the worst possible health condition and 100 indicating the best possible health condition.

OTHER OUTCOMES:
Sleep latency | From baseline to week 24 and from baseline to week 36
  Change in sleep latency, measured with the Pittsburgh Sleep Quality Index; sleep latency domain, scored on an 0-3 interval scale, on which 0 is indicating more problems with sleep latency and higher score less problems with sleep latency.
Pain self-efficacy | From baseline to week 24 and from baseline to week 36
  Change in pain self-efficacy, measured with the Pain Self-Efficacy Questionnaire, consisting of 10 items from 0 to 6 yielding a total score from 0 to 60. Lower scores are indicating lower levels of pain self-efficacy and higher scores are indicating higher levels of pain self-efficacy.
Stiffness | From baseline to week 24 and from baseline to week 36
  Change in stiffness, measured with the Fibromyalgia Impact Questionnaire Revised; stiffness subscale, which is an 11- point numieric rating scale of 0-10, with 10 being the worst outcome indicating the highest level of stiffness, and lower scores indicating less stiffness.
Energy level | From baseline to week 24 and from baseline to week 36
  Change in energy, measured with the Fibromyalgia Impact Questionnaire Revised; energy subscale, which is an 11- point numeric rating scale of 0-10, with10 being the worst outcome, indicating the lowest level of energy, and lower scores indicating higher levels of energy.
Objectively measured physical activity | From baseline to week 24
  Change in objectively measured physical activity, measured with the Sens triaxial accelerometer device; MOTION® activity and sleep measurement system, in which the number of minutes of physical activity are calculated during a week of measurement.
Feeling rested | From baseline to week 24 and from baseline to week 36
  Change in feeling rested, measured with the Fibromyalgia Impact Questionnaire Revised; rested subscale, which is an 11- point numeric rating scale of 0-10, with 10 being the worst outcome indicating not feeling rested, and lower scores indicating feeling more rested.
Depression | From baseline to week 24 and from baseline to week 36
  Change in depression, measured with the Fibromyalgia Impact Questionnaire Revised; depression subscale, which is an 11- point numeric rating scale of 0-10, with 10 being the worst outcome indicating depression, and lower scores indicating less depression, and the Depression, Anxiety, Stress Scale (DASS), depression subscales, which include 7 items scored from 0 to 3 to a maximum of 21 indicating the worst outcome as higher scores indicate more depression and lower scores less depression.
Anxiety | From baseline to week 24 and from baseline to week 36
  Change in anxiety, measured with the Fibromyalgia Impact Questionnaire Revised; anxiety subscale, which is an 11- point numeric rating scale of 0-10, with 10 being the worst outcome indicating more anxiety, and lower scores indicating less anxiety, and the Depression, Anxiety, Stress Scale (DASS), anxiety subscales, which include 7 items scored from 0 to 3 to a maximum of 21 indicating the worst outcome as higher scores indicate more anxiety and lower scores less anxiety.
Perceived stress | From baseline to week 24 and from baseline to week 36
  Change in perceived stress, measured with the Fibromyalgia Impact Questionnaire Revised; stress subscale, which is an 11- point numeric rating scale of 0-10, with 10 being the worst outcome indicating more stress, and lower scores indicating less stress, and the Depression, Anxiety, Stress Scale (DASS), stress subscales, which include 7 items scored from 0 to 3 to a maximum of 21 indicating the worst outcome as higher scores indicate more stress and lower scores less stress.
Cortisol concentration in hair | From baseline to week 24
  Change in cortisol concentration in hair, with hair clipping analysis as a biomarker for prolonged stress. Higher cortisol concentration in hair is indicating higher stress levels.
Memory problems | From baseline to week 24 and from baseline to week 36
  Change in memory problems, measured with the Fibromyalgia Impact Questionnaire Revised; memory subscale, which is an 11- point numeric rating scale of 0-10, with 10 being the worst outcome indicating more memory problems, and lower scores indicating less memory problems.
Tenderness level | From baseline to week 24 and from baseline to week 36
  Change in tenderness level, measured with the Fibromyalgia Impact Questionnaire Revised; tenderness subscale, which is an 11- point numeric rating scale of 0-10, with 10 being the worst outcome indicating more tenderness, and lower scores indicating less tenderness.
Balance problems | From baseline to week 24 and from baseline to week 36
  Change in balance problems, measured with the Fibromyalgia Impact Questionnaire Revised; balance subscale, which is an 11- point numeric rating scale of 0-10, with 10 being the worst outcome indicating more balance problems, and lower scores indicating less balance problems.
Environmental sensitivity | From baseline to week 24 and from baseline to week 36
  Change in environmental sensitivity, measured with the Fibromyalgia Impact Questionnaire Revised; environmental sensitivity subscale, which is an 11- point numeric rating scale of 0-10, with 10 being the worst outcome indicating more environmental sensitivity, and lower scores indicating less environmental sensitivity, and the Fibromyalgia Sensory Hypersensitivity Scale, which is 9 item scale ranging from 0-3 with the maximum score of 27 being the worst outcome indicating the highest level of environmental sensitivity and lower levels indicating less environmental sensitivity.
Pressure pain threshold and tolerance | From baseline to week 24
  Change in pressure pain threshold and tolerance, measured with computerized cuff pressure algometry. Pain threshold is defined as the pressure of the cuff at the subjects first sensation of pain when applying constantly rising pressure. Pain tolerance is defined as the worst tolerable pain caused by the pressure stimulation and the pressure is switched off by the patient. Lower pressures indicates low pressure pain threshold and tolerance, and higher pressures indicates higher pain threshold and tolerance.
Muscle fatiguability | From baseline to week 24
  Change in muscle fatiguability, measured with a static muscle exhaustion test performed during which surface electromyography is recorded. The more muscle exhaustion detected, the more muscle fatiguability.
Appetite | From baseline to week 24 and from baseline to week 36
  Change in appetite, measured with the Simplified Nutritional Appetite Questionnaire, which is a 5 item scale each ranging from 1 to 5, yielding a maximun score of 25. Higher scores are indicating a greater appetite and lower scores are indicating reduced appetite.
Body weight | From baseline to week 24 and from baseline to week 36
  Change in body weight, measured using an electronic scale.
Body composition | From baseline to week 24
  Change in body composition, measured by the bioimpedance measurement conducted using the device named Impedimed model Sfb7, which measures impedance (resistance) through weak electric current flowing through body tissues over a spectrum of frequencies, to detect different body compositions such as body fat and muscle mass, total body water and fat free body mass.
Waist circumference | From baseline to week 24
  Change in waist circumference, will be measured using a tape measure to the nearest 0.1 cm. as a measure of body fat distribution.
Hip circumference | From baseline to week 24
  Change in hip circumference, will be measured using a tape measure to the nearest 0.1 cm. as a measure of body fat distribution.
Pain intensity | From baseline to week 36
  Change in pain intensity, measured with the 0-10 pain Numeric Rating Scale (NRS) item from the Fibromyalgia Impact Questionnaire Revised. The minimum value is 0, which is the best outcome, indicating no pain. The maximum value is 10, which is the worst outcome, indicating the worst possible pain.
Sleep quality | From baseline to week 36
  Change in sleep quality, measured with the Pittsburgh Sleep Quality Index; total score to measure overall sleep quality. Scores are ranging from 0 to 21, with lower scores indictating a better sleep quality and higher scores a worse sleep quality.
Sleep duration | From baseline to week 36
  Change in sleep duration, measured with the Pittsburgh Sleep Quality Index; sleep duration domain, with number of hours of actual sleep during the night.
Activities of daily living | From baseline to week 36
  Change in activities of daily living, measured with the Activities of Daily Living Questionnaire, in which items are rated on a 4 point Likert scale from 0= no problem to 3=no longer able to complete the task. Scores are calculated for total and subscale scores and expressed as a percentage from 0 to 100%. A lower scores percentage indicates a higher level of ADL, and higher percentage indicates a lower level of ADL.
Health-related quality of life | From baseline to week 36
  Change in quality of life, measured with the EuroQol Self-Rated Health Questionnaire, developed by the EuroQual group and international network of multidisciplinary researchers.The scores goes from 0 -100, with 0 indicating the worst possible health condition and 100 indicating the best possible health condition.

CONTACTS AND LOCATIONS:
Overall Officials: Kirstine Amris, Dr. Med, Principal Investigator — The Parker Institute, Frederiksberg University Hospital, Copenhagen, Denmark
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jones GT, Atzeni F, Beasley M, Fluss E, Sarzi-Puttini P, Macfarlane GJ. The prevalence of fibromyalgia in the general population: a comparison of the American College of Rheumatology 1990, 2010, and modified 2010 classification criteria. Arthritis Rheumatol. 2015 Feb;67(2):568-75. doi: 10.1002/art.38905. PMID 25323744
- [Background] Walitt B, Nahin RL, Katz RS, Bergman MJ, Wolfe F. The Prevalence and Characteristics of Fibromyalgia in the 2012 National Health Interview Survey. PLoS One. 2015 Sep 17;10(9):e0138024. doi: 10.1371/journal.pone.0138024. eCollection 2015. PMID 26379048
- [Background] Wolfe F, Brahler E, Hinz A, Hauser W. Fibromyalgia prevalence, somatic symptom reporting, and the dimensionality of polysymptomatic distress: results from a survey of the general population. Arthritis Care Res (Hoboken). 2013 May;65(5):777-85. doi: 10.1002/acr.21931. PMID 23424058
- [Background] Smith HS, Harris R, Clauw D. Fibromyalgia: an afferent processing disorder leading to a complex pain generalized syndrome. Pain Physician. 2011 Mar-Apr;14(2):E217-45. PMID 21412381
- [Background] Coster L, Kendall S, Gerdle B, Henriksson C, Henriksson KG, Bengtsson A. Chronic widespread musculoskeletal pain - a comparison of those who meet criteria for fibromyalgia and those who do not. Eur J Pain. 2008 Jul;12(5):600-10. doi: 10.1016/j.ejpain.2007.10.001. Epub 2007 Nov 19. PMID 18024204
- [Background] Hallberg LR, Carlsson SG. Coping with fibromyalgia. A qualitative study. Scand J Caring Sci. 2000;14(1):29-36. doi: 10.1111/j.1471-6712.2000.tb00558.x. PMID 12035259
- [Background] Bandak E, Amris K, Bliddal H, Danneskiold-Samsoe B, Henriksen M. Muscle fatigue in fibromyalgia is in the brain, not in the muscles: a case-control study of perceived versus objective muscle fatigue. Ann Rheum Dis. 2013 Jun;72(6):963-6. doi: 10.1136/annrheumdis-2012-202340. Epub 2012 Dec 8. PMID 23223425
- [Background] Amris K, Waehrens EE, Jespersen A, Bliddal H, Danneskiold-Samsoe B. Observation-based assessment of functional ability in patients with chronic widespread pain: a cross-sectional study. Pain. 2011 Nov;152(11):2470-2476. doi: 10.1016/j.pain.2011.05.027. Epub 2011 Jun 28. PMID 21715094
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Sjogren P, Ekholm O, Peuckmann V, Gronbaek M. Epidemiology of chronic pain in Denmark: an update. Eur J Pain. 2009 Mar;13(3):287-92. doi: 10.1016/j.ejpain.2008.04.007. Epub 2008 Jun 10. PMID 18547844
- [Background] Ablin JN, Buskila D. Emerging therapies for fibromyalgia: an update. Expert Opin Emerg Drugs. 2010 Sep;15(3):521-33. doi: 10.1517/14728214.2010.491509. PMID 20486862
- [Background] Hauser W, Walitt B, Fitzcharles MA, Sommer C. Review of pharmacological therapies in fibromyalgia syndrome. Arthritis Res Ther. 2014 Jan 17;16(1):201. doi: 10.1186/ar4441. PMID 24433463
- [Background] Smith HS, Bracken D, Smith JM. Pharmacotherapy for fibromyalgia. Front Pharmacol. 2011 Mar 31;2:17. doi: 10.3389/fphar.2011.00017. eCollection 2011. PMID 21772818
- [Background] Hauser W, Wolfe F, Tolle T, Uceyler N, Sommer C. The role of antidepressants in the management of fibromyalgia syndrome: a systematic review and meta-analysis. CNS Drugs. 2012 Apr 1;26(4):297-307. doi: 10.2165/11598970-000000000-00000. PMID 22452526
- [Background] Hauser W, Urrutia G, Tort S, Uceyler N, Walitt B. Serotonin and noradrenaline reuptake inhibitors (SNRIs) for fibromyalgia syndrome. Cochrane Database Syst Rev. 2013 Jan 31;(1):CD010292. doi: 10.1002/14651858.CD010292. PMID 23440848
- [Background] Moore RA, Straube S, Wiffen PJ, Derry S, McQuay HJ. Pregabalin for acute and chronic pain in adults. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD007076. doi: 10.1002/14651858.CD007076.pub2. PMID 19588419
- [Background] Moore RA, Derry S, Aldington D, Cole P, Wiffen PJ. Amitriptyline for neuropathic pain and fibromyalgia in adults. Cochrane Database Syst Rev. 2012 Dec 12;12:CD008242. doi: 10.1002/14651858.CD008242.pub2. PMID 23235657
- [Background] Tort S, Urrutia G, Nishishinya MB, Walitt B. Monoamine oxidase inhibitors (MAOIs) for fibromyalgia syndrome. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD009807. doi: 10.1002/14651858.CD009807. PMID 22513976
- [Background] Uceyler N, Sommer C, Walitt B, Hauser W. Anticonvulsants for fibromyalgia. Cochrane Database Syst Rev. 2013 Oct 16;(10):CD010782. doi: 10.1002/14651858.CD010782. PMID 24129853
- [Background] Wiffen PJ, Derry S, Moore RA, Aldington D, Cole P, Rice AS, Lunn MP, Hamunen K, Haanpaa M, Kalso EA. Antiepileptic drugs for neuropathic pain and fibromyalgia - an overview of Cochrane reviews. Cochrane Database Syst Rev. 2013 Nov 11;2013(11):CD010567. doi: 10.1002/14651858.CD010567.pub2. PMID 24217986
- [Background] Moore AR, Straube S, Paine J, Phillips CJ, Derry S, McQuay HJ. Fibromyalgia: Moderate and substantial pain intensity reduction predicts improvement in other outcomes and substantial quality of life gain. Pain. 2010 May;149(2):360-364. doi: 10.1016/j.pain.2010.02.039. Epub 2010 Mar 26. PMID 20347225
- [Background] Ste-Marie PA, Fitzcharles MA, Gamsa A, Ware MA, Shir Y. Association of herbal cannabis use with negative psychosocial parameters in patients with fibromyalgia. Arthritis Care Res (Hoboken). 2012 Aug;64(8):1202-8. doi: 10.1002/acr.21732. PMID 22730275
- [Background] Lynch ME, Campbell F. Cannabinoids for treatment of chronic non-cancer pain; a systematic review of randomized trials. Br J Clin Pharmacol. 2011 Nov;72(5):735-44. doi: 10.1111/j.1365-2125.2011.03970.x. PMID 21426373
- [Background] Bramness JG, Dom G, Gual A, Mann K, Wurst FM. A Survey on the Medical Use of Cannabis in Europe: A Position Paper. Eur Addict Res. 2018;24(4):201-205. doi: 10.1159/000492757. Epub 2018 Aug 22. PMID 30134238
- [Background] Pertwee RG. The diverse CB1 and CB2 receptor pharmacology of three plant cannabinoids: delta9-tetrahydrocannabinol, cannabidiol and delta9-tetrahydrocannabivarin. Br J Pharmacol. 2008 Jan;153(2):199-215. doi: 10.1038/sj.bjp.0707442. Epub 2007 Sep 10. PMID 17828291
- [Background] Iffland K, Grotenhermen F. An Update on Safety and Side Effects of Cannabidiol: A Review of Clinical Data and Relevant Animal Studies. Cannabis Cannabinoid Res. 2017 Jun 1;2(1):139-154. doi: 10.1089/can.2016.0034. eCollection 2017. PMID 28861514
- [Background] Millar SA, Stone NL, Yates AS, O'Sullivan SE. A Systematic Review on the Pharmacokinetics of Cannabidiol in Humans. Front Pharmacol. 2018 Nov 26;9:1365. doi: 10.3389/fphar.2018.01365. eCollection 2018. PMID 30534073
- [Background] Morales P, Hernandez-Folgado L, Goya P, Jagerovic N. Cannabinoid receptor 2 (CB2) agonists and antagonists: a patent update. Expert Opin Ther Pat. 2016 Jul;26(7):843-56. doi: 10.1080/13543776.2016.1193157. Epub 2016 Jun 7. PMID 27215781
- [Background] Temple LM. Medical marijuana and pain management. Dis Mon. 2016 Sep;62(9):346-52. doi: 10.1016/j.disamonth.2016.05.014. Epub 2016 Jun 27. No abstract available. PMID 27364691
- [Background] Wise J. FDA approves its first cannabis based medicine. BMJ. 2018 Jun 27;361:k2827. doi: 10.1136/bmj.k2827. No abstract available. PMID 29950322
- [Background] Drug Enforcement Administration, Department of Justice. Schedules of Controlled Substances: Placement of FDA-Approved Products of Oral Solutions Containing Dronabinol [(-)-delta-9-transtetrahydrocannabinol (delta-9-THC)] in Schedule II. Interim final rule, with request for comments. Fed Regist. 2017 Mar 23;82(55):14815-20. PMID 28355049
- [Background] Bifulco M, Pisanti S. Medicinal use of cannabis in Europe: the fact that more countries legalize the medicinal use of cannabis should not become an argument for unfettered and uncontrolled use. EMBO Rep. 2015 Feb;16(2):130-2. doi: 10.15252/embr.201439742. Epub 2015 Jan 9. No abstract available. PMID 25576303
- [Background] Walitt B, Klose P, Fitzcharles MA, Phillips T, Hauser W. Cannabinoids for fibromyalgia. Cochrane Database Syst Rev. 2016 Jul 18;7(7):CD011694. doi: 10.1002/14651858.CD011694.pub2. PMID 27428009
- [Background] Stockings E, Campbell G, Hall WD, Nielsen S, Zagic D, Rahman R, Murnion B, Farrell M, Weier M, Degenhardt L. Cannabis and cannabinoids for the treatment of people with chronic noncancer pain conditions: a systematic review and meta-analysis of controlled and observational studies. Pain. 2018 Oct;159(10):1932-1954. doi: 10.1097/j.pain.0000000000001293. PMID 29847469
- [Background] Fiz J, Duran M, Capella D, Carbonell J, Farre M. Cannabis use in patients with fibromyalgia: effect on symptoms relief and health-related quality of life. PLoS One. 2011 Apr 21;6(4):e18440. doi: 10.1371/journal.pone.0018440. PMID 21533029
- [Background] Piper BJ, Beals ML, Abess AT, Nichols SD, Martin MW, Cobb CM, DeKeuster RM. Chronic pain patients' perspectives of medical cannabis. Pain. 2017 Jul;158(7):1373-1379. doi: 10.1097/j.pain.0000000000000899. PMID 28328576
- [Background] Habib G, Artul S. Medical Cannabis for the Treatment of Fibromyalgia. J Clin Rheumatol. 2018 Aug;24(5):255-258. doi: 10.1097/RHU.0000000000000702. PMID 29461346
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Choy EH, Arnold LM, Clauw DJ, Crofford LJ, Glass JM, Simon LS, Martin SA, Strand CV, Williams DA, Mease PJ. Content and criterion validity of the preliminary core dataset for clinical trials in fibromyalgia syndrome. J Rheumatol. 2009 Oct;36(10):2330-4. doi: 10.3899/jrheum.090368. PMID 19820222
- [Background] Bennett RM, Friend R, Jones KD, Ward R, Han BK, Ross RL. The Revised Fibromyalgia Impact Questionnaire (FIQR): validation and psychometric properties. Arthritis Res Ther. 2009;11(4):R120. doi: 10.1186/ar2783. Epub 2009 Aug 10. PMID 19664287
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Background] Waehrens EE, Bliddal H, Danneskiold-Samsoe B, Lund H, Fisher AG. Differences between questionnaire- and interview-based measures of activities of daily living (ADL) ability and their association with observed ADL ability in women with rheumatoid arthritis, knee osteoarthritis, and fibromyalgia. Scand J Rheumatol. 2012 Mar;41(2):95-102. doi: 10.3109/03009742.2011.632380. Epub 2012 Jan 30. PMID 22283877
- [Background] Nicholas MK. The pain self-efficacy questionnaire: Taking pain into account. Eur J Pain. 2007 Feb;11(2):153-63. doi: 10.1016/j.ejpain.2005.12.008. Epub 2006 Jan 30. PMID 16446108
- [Background] Rasmussen MU, Rydahl-Hansen S, Amris K, Samsoe BD, Mortensen EL. The adaptation of a Danish version of the Pain Self-Efficacy Questionnaire: reliability and construct validity in a population of patients with fibromyalgia in Denmark. Scand J Caring Sci. 2016 Mar;30(1):202-10. doi: 10.1111/scs.12232. Epub 2015 Apr 29. PMID 25924021
- [Background] Henry JD, Crawford JR. The short-form version of the Depression Anxiety Stress Scales (DASS-21): construct validity and normative data in a large non-clinical sample. Br J Clin Psychol. 2005 Jun;44(Pt 2):227-39. doi: 10.1348/014466505X29657. PMID 16004657
- [Background] Nielsen MG, Ornbol E, Vestergaard M, Bech P, Larsen FB, Lasgaard M, Christensen KS. The construct validity of the Perceived Stress Scale. J Psychosom Res. 2016 May;84:22-30. doi: 10.1016/j.jpsychores.2016.03.009. Epub 2016 Mar 16. PMID 27095155
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Wilson MM, Thomas DR, Rubenstein LZ, Chibnall JT, Anderson S, Baxi A, Diebold MR, Morley JE. Appetite assessment: simple appetite questionnaire predicts weight loss in community-dwelling adults and nursing home residents. Am J Clin Nutr. 2005 Nov;82(5):1074-81. doi: 10.1093/ajcn/82.5.1074. PMID 16280441
- [Background] Jespersen A, Dreyer L, Kendall S, Graven-Nielsen T, Arendt-Nielsen L, Bliddal H, Danneskiold-Samsoe B. Computerized cuff pressure algometry: A new method to assess deep-tissue hypersensitivity in fibromyalgia. Pain. 2007 Sep;131(1-2):57-62. doi: 10.1016/j.pain.2006.12.012. Epub 2007 Jan 25. PMID 17257757
- [Background] Van Uum SH, Sauve B, Fraser LA, Morley-Forster P, Paul TL, Koren G. Elevated content of cortisol in hair of patients with severe chronic pain: a novel biomarker for stress. Stress. 2008 Nov;11(6):483-8. doi: 10.1080/10253890801887388. PMID 18609301
- [Background] Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Dore C, Williamson PR, Altman DG, Montgomery A, Lim P, Berlin J, Senn S, Day S, Barbachano Y, Loder E. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. JAMA. 2017 Dec 19;318(23):2337-2343. doi: 10.1001/jama.2017.18556. PMID 29260229
- [Background] de Wit MP, Berlo SE, Aanerud GJ, Aletaha D, Bijlsma JW, Croucher L, Da Silva JA, Glusing B, Gossec L, Hewlett S, Jongkees M, Magnusson D, Scholte-Voshaar M, Richards P, Ziegler C, Abma TA. European League Against Rheumatism recommendations for the inclusion of patient representatives in scientific projects. Ann Rheum Dis. 2011 May;70(5):722-6. doi: 10.1136/ard.2010.135129. Epub 2011 Jan 20. PMID 21257615
- [Background] Sundhedsstyrelsen, Callesen H, von Bülow C, Birkefoss K, Rasmussen M (2018) Nationale kliniske retningslinjer for udredning og behandling samt rehabilitering af patienter med genrelaliserede smerter i bevægeapparatet. https://www.sst.dk/da/udgivelser/2018/~/media/82268C6BAF19461399C4FC8D1647DCC0.ashx.
- [Background] Lov om forsøgsordning med medicinsk cannabis. https://www.retsinformation.dk/Forms/R0710.aspx?id=196748 (2018).
- [Background] Nabilone. https://pubchem.ncbi.nlm.nih.gov/compound/Nabilone#section=Top (2018)
- [Background] Banerjee S, McCormack S. Medical Cannabis for the Treatment of Chronic Pain: A Review of Clinical Effectiveness and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2019 Jul 24. Available from http://www.ncbi.nlm.nih.gov/books/NBK546424/ PMID 31532599
- [Background] Fisher, A. G. (2010) Assessment of Motor and Process Skills: Development, Standardization, and Administration Manual. Fort Collins, Colorado: Three Star Press.
- [Background] Sens Motion (2020) Discrete Wearable Acticity Sensor for Healthcare and Research.
- [Background] ImpediMed, SFB7 (2020) ImpediMed.
- [Background] Pro.medicin Information til sundhedsfaglige (2018) Sativex. https://pro.medicin.dk/Medicin/Praeparater/6456.
- [Background] Greenwich Biosciences I (2020) Epidiolex Highlights of Prescibing Information.
- [Background] (2020) Epidyolex Summary of product characteristics.
- [Derived] Rasmussen MU, Christensen R, Waehrens EE, Henriksen M, Duhn PH, Bliddal H, Amris K. Cannabidiol versus placebo in patients with fibromyalgia: a randomised, double-blind, placebo-controlled, parallel-group, single-centre trial. Ann Rheum Dis. 2025 Aug 21:S0003-4967(25)04238-4. doi: 10.1016/j.ard.2025.07.008. Online ahead of print. PMID 40846590

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Protocol only (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT04729179/Prot_SAP_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Pan (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04729179/SAP_001.pdf